CLINICAL TRIAL: NCT06225323
Title: Effect of Lidocaine Infusion on Neuraxial Opioid-induced Pruritus After Cesarean Section Double-blinded, Randomized Control Clinical Trial
Brief Title: Effect of Lidocaine Infusion on Neuraxial Opioid-induced Pruritus After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Ayman Mohamady Eldemrdash, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Aswu/668/10/22
Record Dates: First submitted 2024-01-17; First posted 2024-01-25 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Lidocaine Infusion; Neuraxial Opioid; Pruritus; Cesarean Section
MeSH Terms: conditions — Pruritus | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Patients will receive Lidocaine infusion for 6 hours
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): Patients will receive normal saline infusion for 6 hours
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Lidocaine — Patients will receive Lidocaine infusion for 6 hours. After cord clamping and according to ideal body calculate the bolus dose 1.5 mg/kg of lidocaine 1% and complete the dose by normal saline to 20 ml total volume will be given in 10 min.
  The infusion dose 1.5 mg/kg/hour of lidocaine 1% for 6 hours in automated syringe pump (aquavesar fixed variable rate 100ml volume) 100 ml then follow up without infusion up to 24 hours.
  Arms: Lidocaine group
Other: Saline — Patients will receive normal saline infusion for 6 hours. After cord clamping 20 ml total volume normal saline will be given in 10 min.
  The infusion dose 1.5 mg/kg/hour of normal saline for 6 hours in automated syringe pump (aquavesar fixed variable rate 100ml volume) 100 ml then follow up without infusion up to 24 hours.
  Arms: Control group

SUMMARY:
The aim of this study is to assess the efficacy and potency of lidocaine infusion as a preventive measure on pruritus response after injection of 200 micro gram morphine with bupivacaine subarachnoid block, spinal anesthesia, in cesarean section.

DETAILED DESCRIPTION:
Neuraxial opioids (NO) are one of the most widely used methods for postpartum analgesia, for cesarean section analgesia, and many other surgical procedures.

The pruritus induced by NO is an unpleasant, subjective, and irritating sensation that causes scratching response.

Pruritus begins shortly after anesthesia, with the onset depending on the type, route and dosage of opioid used. Pruritus invoked by lipid-soluble opioids such as fentanyl and sufentanil is of shorter duration, and the use of the minimum or small dose from opioids in addition of local anesthetics seems to decrease the prevalence and the severity of itching. Pruritus invoked by intrathecal morphine is of longer duration and is difficult to treat. Intrathecal administration, of opioids reach peak concentrations in the cerebrospinal fluid almost immediately. ]. But, after epidural administration, there is a delay in the rise to peak concentration (10-20 min with fentanyl and 1-4 h with morphine).

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 40 years.
* Weight from 50 to 90 kg.
* Women undergoing Cesarean section.

Exclusion Criteria:

* Patient with known allergies to lidocaine.
* Preexisting pruritus.
* Coexisting skin disorders.
* Contraindications to spinal anesthesia.
* Preeclampsia.
* Eclampsia.
* Major systemic diseases.
* Refusal to participate.
* Uses of any current drugs have potential effects on post-operative itching as steroidal ,nonsteroidal ,ondanstern, propofol, midazolam during study period.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing Cesarean section
Enrollment: 136 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The incidence of pruritis | 24 hours postoperatively
  The incidence of pruritis will be classifies as moderate (affecting a larger area, such as face and arms or face and anterior surface of thorax, but not disturbing the patient, and therefore not requiring treatment) , severe (extensive or generalized, often disturbing the patient and may need treatment)or very sever(disturbing the patient and treatment was indicated).

SECONDARY OUTCOMES:
The severity of pruritis | 24 hours postoperatively
  The severity of pruritis will be assessed using qualitative scales (Pruritus Severity Scale)such as none, mild, moderate, severe or very sever pruritus.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.